CLINICAL TRIAL: NCT03061409
Title: Vitamin and Mineral Supplementation Improves Micronutrient Status in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: MB Clinical Research and Consulting LLC (Unknown)
Responsible Party: Principal Investigator, Jeffrey Blumberg, Research Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2900
Record Dates: First submitted 2017-01-12; First posted 2017-02-23 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Nutrient Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmavite Nature Made Multi for Him 50+ (Experimental): A supplement containing vitamins and minerals
  Interventions: Dietary Supplement: Pharmavite Nature Made Multi for Him 50+
- placebo (Placebo Comparator): tablets contain microcrystalline cellulose containing 0.5% magnesium stearate
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pharmavite Nature Made Multi for Him 50+ — To examine whether one tablet a day of Pharmavite Nature Made Multi for Him 50+ will increase micro-nutrient status in older people taking multiple medications as compared to placebo
  Arms: Pharmavite Nature Made Multi for Him 50+
Dietary Supplement: Placebo — served as placebo
  Arms: placebo

SUMMARY:
Nutrient intake through diet and nutritional supplements are critical determinants of plasma nutrient status. In addition, untoward drug-nutrient can contribute to nutritional inadequacy. Among medications used by the elderly in the US, diuretics, metformin, and proton pump inhibitors (PPIs) are ranked among the most commonly prescribed. Use of these medications is variously associated with inadequate status of many micronutrients, e.g., vitamins B1, B9 (folate), B12, C, and thiamine and the minerals calcium, iron, potassium, magnesium, and zinc. While diets rich in whole grains, fruits, and vegetables can help decrease the risk for micronutrient inadequacy in older adults using one or more of these drugs, supplementation may prove more effective to restoring and/or enhancing their nutrient status. When compared to a placebo, investigators hypothesize that a multivitamin-multi-mineral (MVM) supplement will improve nutritional status in older adults at increased risk of micronutrient inadequacy induced by drugs commonly used by this population, specifically diuretics, metformin, and PPIs. Investigators also hypothesize that MVM supplementation will beneficially modify selected biomarkers or biochemical pathways of cellular function/health. To test these hypotheses, investigators will conduct a randomized clinical trial by pursuing the following specific aims: 1) To determine the extent by which MVM supplementation (compared to placebo) will increase the plasma status of vitamins B12, C, D, folic acid, and thiamine and the minerals iron, magnesium, potassium, and zinc; 2) To quantify indices of 'metabolic health' including one or more of the following biomarkers: glutathione (GSH)/glutathione disulfide (GSSG) ratio, ubiquinol/ubiquinone, malondialdehyde (MDA), asymmetric dimethyl arginine (ADMA), selected cytokines and chemokines, homocysteine, methylmalonic acid (MMA).

DETAILED DESCRIPTION:
The older adults are prone to inadequate nutrition. The prevalence of malnutrition is 5-10% among independently living older individuals, 30-60% among institutionalized patients, and 35-65% among hospitalized geriatric patients. There are many factors that make the elderly more susceptible to nutrition inadequacy. Aging itself is associated with a decline in a number of physiological functions that can impact nutritional status, including reduced lean body mass and a resultant decrease in basal metabolic rate, decreased gastric secretion of digestive juices and changes in the oral cavity, sensory function deficits, changes in fluid and electrolyte regulation, and chronic diseases. In addition, medications can contribute to nutritional inadequacy through many mechanisms, from decreased nutrient absorption in the gastrointestinal tract to increased metabolism and from enhanced utilization to rapid elimination It has been reported there are >250 drugs that may influence the intake, absorption, metabolism and excretion of nutrients. As Americans rely more on prescription drugs, many are taking multiple drugs daily, so polypharmacy can increase the likelihood of drug-nutrition interactions through additive and synergistic actions.

Investigators will conduct a randomized, double-blind, placebo controlled, parallel clinical trial to test the hypotheis. This trial will include 72 older adults randomized to receive either placebo or MVM supplement. Participants will be 45-75 y and have a BMI >20 and <36 kg/m2. Participants will be receiving regular, chronic pharmacotherapy with ≥2 drugs in the following drug classes: a diuretic, metformin and/or proton pump inhibitor medication with allowance for a total of less than 7 drug prescriptions. The medication history with one of the target drugs will be longer than 6 mo. The total duration of the trial will be ~5 mo, including screening and 16 wk of intervention. Participants must maintain their medication regimens and dietary habits throughout the intervention. During the intervention phase, Participants will take the assigned supplement daily. Blood and urine samples will be collected at the baseline, 8 wk, and the end of the 16 wk intervention.

Participants will be randomly assigned to receive one of the supplements (MVM vs. placebo) after their eligibility is confirmed. A randomization scheme will be prepared by a biostatistician using a standardized computer program for two treatment groups using a parallel design. The nutrient composition of MVM supplement, which will be Pharmavite Nature Made Multi for Him 50+ (newly manufactured). A matching placebo product will be manufactured by the Natural Alternatives International, Inc. (San Marcos, CA) under the FDA Good Manufacturing Practices(GMP) guidelines. The main ingredient of the placebo will be microcrystalline cellulose containing 0.5% magnesium stearate. Pharmavite Nature Made Multi for Him 50+ has been marketed in US, and both microcrystalline cellulose and magnesium stearate have a Generally Recognized As Safe (GRAS) status under FDA Code of Federal Regulations (CFR) title 21.

ELIGIBILITY:
Inclusion Criteria:

1. BMI, 20-36 kg/m2
2. Taking two or more of the following prescribed drugs (with allowance for a total of more than 6 drug prescriptions):

   1. diuretic, including: Thiazides: chlorothiazide (Diuril), hydrochlorothiazide (Hydrodiuril), indapamide (Lozol), metolazone (Zaroxolyn), chlorthalidone (Hygroton), methyclothiazide (Enduron); Potassium-sparing: amiloride hydrochloride, spironolactone (Aldactone), triamterene (Dyrenium); Loop: bumetanide (Bumex), furosemide (Lasix), ethacrynate (Edecrin), torsemide (Demadex); and Carbonic anhydrase inhibitors: acetazolamide, methazolamide
   2. metformin, including: Fortamet, Glucophage, Glumetza, Riomet, ActoPlus Met (with pioglitazone), Avandamet (with rosiglitazone), Glucovance (with glyburide), Janumet (with sitagliptin), Jentadueto (with linagliptin), Kombiglyze extended release (with saxagliptin), Invokamet (with canagliflozin), Metaglip (with glipizide), and PrandiMet (with repaglinide)
   3. PPI, including: dexlansoprazole (Dexilant, Kapidex), esomeprazole (Nexium) lansoprazole (Prevacid), omeprazole (Prilosec, Zegarid), pantoprazole (Protonix), and rabeprazole (Aciphex)]
3. Willing to take the assigned supplement for 16 wk.
4. Willing to maintain dietary habit for 16 wk.

Exclusion Criteria:

1. Unusual dietary pattern, including vegan/vegetarian.
2. Pregnant or intend to be pregnant.
3. Active treatment for cancer of any type longer than 1 y.
4. Daily alcoholic intake of more than 14 drinks/wk (168 oz beer, 56 oz wine, 14 oz hard liquor).
5. Regular use of any dietary supplements containing vitamins and minerals; however, subjects who are willing to refrain from the use of these supplements for 1 mo prior to their enrollment and throughout the entire study may be considered eligible; subjects will be excluded if they are taking physician prescribed vitamin and/or mineral supplements (This information will be self reported by subjects and documented in the study record of each subject.).
6. Values of standard blood biochemistries are critically abnormal based on study physician's discretion.
7. Taking >6 prescription or over-the-counter (OTC) drugs on a chronic basis.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline nutrient status at 16 weeks | 0 and 16 weeks
  Vitamin B6, B12, folic acid, thiamine, calcium, magnesium, zinc in plasma will be qunantified.

SECONDARY OUTCOMES:
Change from Baseline redox status at 16 weeks | 0 and 16 weeks
  plasma biomarkers of free radical attacked products will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Blumberg, PhD, Principal Investigator — Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging, Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No